CLINICAL TRIAL: NCT06532162
Title: The PRICE Trial: Pain Reduction for Intrauterine Contraception Experiment. a Double-blind, Triple Arm, Randomized Controlled Trial of 1% Lidocaine Paracervical Block for IUD Insertion
Brief Title: The PRICE Trial: Pain Reduction for Intrauterine Contraception Experiment
Acronym: PRICE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mount Sinai Hospital, Canada (Other)
Responsible Party: Principal Investigator, Mara Sobel, Associate Professor, Mount Sinai Hospital, Canada
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PRICE Trial
Record Dates: First submitted 2024-07-29; First posted 2024-08-01 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Contraception
Keywords: Contraception; Intrauterine device; Paracervical block

STUDY DESIGN:
Intervention Model Description: The proposed study is a double-blind, triple arm, placebo-controlled randomized clinical trial. Participants will be recruited from Mount Sinai Hospital outpatient gynecology clinics. Recruitment, consent, randomization, procedure, and post-procedure survey will occur during the same visit. Each participant will be randomly assigned to one of three arms:
  1. Intervention (10 cc 1% lidocaine paracervical block)
  2. Placebo (10 cc paracervical injection of normal saline)
  3. Control (gently tapping the cervicovaginal junction with a capped needle)
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: We will employ two providers to ensure a double-blinded set-up. The first provider (Provider A) will open the allocation envelopes without the presence of the participant or second provider (Provider B).
  Provider A will then enter the patient's room and introduce themselves. They will place the speculum, and administer either the intervention, placebo, or control and then leave the room after injection-related bleeding has stopped. After 3 minutes, the second provider (Provider B) will enter the room to place the IUD (including sounding and tenaculum placement) and will be unaware of the participant's treatment arm.
  A standardized script will be used with all participants: "You may or not may feel a poke."
  Both lidocaine and the control (normal saline) are odorless and clear, minimizing the risk of unblinding. All data will remain blinded until data analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- 1% Lidocaine Paracervical Block (Experimental): A 22-gauge spinal needle will be loaded with 10 mL of 1% lidocaine with epinephrine.
  The injection will be instilled slowly over 60 seconds into the cervicovaginal junction in two equal areas at 2 and 10 o'clock. The injection is continuous from superficial to deep (3 cm).
  Interventions: Drug: 1% Lidocaine Paracervical Block
- Normal Saline Paracervical Injection (Sham Comparator): A 22-gauge spinal needle will be loaded with 10 mL of normal saline. The injection will be instilled slowly over 60 seconds into the cervicovaginal junction in two equal areas at 2 and 10 o'clock. The injection is continuous from superficial to deep (3 cm).
  Interventions: Drug: Normal Saline Paracervical Injection
- Capped Needle Control (No Intervention): A capped needle will gently be tapped on the cervicovaginal junction at two areas at 2 and 10 o'clock.

INTERVENTIONS:
Drug: 1% Lidocaine Paracervical Block — A 22-gauge spinal needle will be loaded with 10 mL of 1% lidocaine with epinephrine.
  The injection will be instilled slowly over 60 seconds into the cervicovaginal junction in two equal areas at 2 and 10 o'clock. The injection is continuous from superficial to deep (3 cm).
  Arms: 1% Lidocaine Paracervical Block
Drug: Normal Saline Paracervical Injection — A 22-gauge spinal needle will be loaded with 10 mL of normal saline. The injection will be instilled slowly over 60 seconds into the cervicovaginal junction in two equal areas at 2 and 10 o'clock. The injection is continuous from superficial to deep (3 cm).
  Arms: Normal Saline Paracervical Injection

SUMMARY:
Intrauterine devices (IUDs) are a highly effective form of reversible contraception with a less than 1% failure rate. They can be easily placed in the office and require little maintenance care. However, despite their benefits, pain during insertion remains a barrier for patient uptake. Currently there is no standard of care for pain management during IUD insertion. The aim of this study is to determine whether local anesthetic, in the form of injecting 1 percent lidocaine into the cervicovaginal junction, reduces pain during insertion. Participants will be randomly assigned to receive 1 percent lidocaine, placebo, or no injection. All patients presenting for IUD placement, regardless of indication, will be offered participation in the study. Following IUD placement, patients will be asked to rate their pain at key "pain points" during the procedure as the primary outcome. Other outcomes collected will include provider-related complications, length of time to place IUD, and overall patient and provider satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Any participant presenting for an IUD placement, either for contraception or treatment of abnormal uterine bleeding or to regulate menstrual periods
* All IUDs (copper, hormonal) eligible
* All parities of patients are eligible

Exclusion Criteria:

* Use of pain medication that is not an NSAID or acetaminophen (e.g. opioids, benzodiazepines) within past 24 hours
* Confirmed pregnancy
* Any diagnosed chronic pain conditions (fibromyalgia, vaginismus, interstitial cystitis)
* Misoprostol administration within 24 hours of enrollment
* Known contraindications to IUD placement
* Contraindication to lidocaine
* IUD exchange
* Previous unsuccessful attempt for IUD by the same practitioner

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 246 (Actual)
Dates: Start 2022-06-30 (Actual); Primary Completion 2024-08-16 (Actual); Study Completion 2024-08-16 (Actual)

PRIMARY OUTCOMES:
Global Pain Score | Immediately following the procedure
  Patient-reported overall pain score on the 100 mm Visual Analogus Scale (VAS). A score of 0 mm is the minimum, 100 mm is the maximum, with higher scores indicating more pain (i.e. worse outcome).

SECONDARY OUTCOMES:
Pain at specific pain points | Baseline, after injection or placebo, tenaculum placement, uterine sounding, IUD insertion, 1 minute post-procedure
  Patient-reported pain score at specific pain points during the procedure, on the 100 mm Visual Analogus Scale (VAS). A score of 0 mm is the minimum, 100 mm is the maximum, with higher scores indicating more pain (i.e. worse outcome).
Immediate complications following the procedure (i.e. vasovagal response, dizziness, local anesthetic toxicity syndrome) | Immediately following the procedure
  Provider reported based on events during the procedure
Length of time for analgesia | Immediately following administration of the intervention, placebo, or control
  Stopwatch
Length of time for IUD placement | Immediately following the procedure
  Stopwatch
Patient satisfaction | Immediately following the procedure
  Survey-related questions, based on Likert scale and yes/no answers
Difficulty of IUD placement | 1 is minimum (least diffiult) and 5 is maximum (most difficult). Higher scores are worse outcome as they are more difficult.
  Provider reported on Likert scale

CONTACTS AND LOCATIONS:
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No